CLINICAL TRIAL: NCT05517096
Title: ALPACA : the Effect of Online Monitoring and Communication on the Quality and Quantity of Pediatric Asthma Care
Brief Title: AmbuLatory Pediatric Asthma CAre
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: refocus of business
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Collaborators: Medisch Spectrum Twente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICBE-S-000177
Record Dates: First submitted 2022-08-18; First posted 2022-08-26 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Asthma in Children
Keywords: E-health

STUDY DESIGN:
Intervention Model Description: In the first phase subjects are block randomized (section 7.2) to either eHealth care and explorative observational home-monitoring or only explorative observational home-monitoring during regular care. The second phase is a follow-up period of 3 months to evaluate the effects of eHealth care compared to the control group and how long these effects can last.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E-Health and monitoring (Experimental): eHealth care and explorative observational home-monitoring
  Interventions: Other: E-Health
- regular care and monitoring (No Intervention): only explorative observational home-monitoring during regular care

INTERVENTIONS:
Other: E-Health — In the intervention phase asthma care is provided on an at-needed-basis via online communication and is always available during working hours.
  Arms: E-Health and monitoring

SUMMARY:
The ALPACA study has a prospective randomized control interventional design, including a follow-up period to evaluate follow-up effects. The study is divided into two phases of 3 months using eHealth and observational monitoring.

DETAILED DESCRIPTION:
The ALPACA study has a prospective randomized control interventional design, including a follow-up period to evaluate follow-up effects. The study is divided into two phases of 3 months; In the first phase subjects are randomized to either eHealth care (use of a communication portal including the weekly entry of SpO2, spirometry results and ACT) and explorative observational home-monitoring or only explorative observational home-monitoring during regular care. The second phase is to evaluate the effects of eHealth care compared to the control group after a follow-up period of 3 months, and the time to healthcare events during follow-up in both groups (survival analysis). The study makes use of an intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children with moderate-to-severe asthma.
* Children in the age group from 4 up to and included 11 years old.

Exclusion Criteria:

* Children living in a house without WIFI.
* Prior participation in eHealth care trial.
* Children/Parents with an inability to understand or speak Dutch.
* Children with divorced parents or other reasons that causes them to be less than 80% on the same living address.
* Children of whom family members have already participated in this trial.
* Children for whom it is not possible to perform at least one of the two discontinuous dyspnea assessment (lung function/pulse oximetry).
* Children using an inhaler that is not compatible with the FindAir smart inhaler cap, which cannot be replaced by a compatible alternative.
* Children with chronic diseases other than asthma (i.e. inflammatory bowel disease, behavioral disorders, mental retardation).
* Currently displaying COVID-19-related symptoms, namely a fever, cough and/or difficulty breathing (during inclusion).
* Having been positively tested as infected with COVID-19 in the past 14 days

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
healthcare utilization | during study period after 6 months
  Difference in utilization of healthcare

SECONDARY OUTCOMES:
assesment of effect of ehealth on asthma outcomes | during study period (3 and 6 months)
  asthma outcome measures
assess the effect of personalized real-time monitoring and education of inhalation | during study period (3 and 6 months)
  monitoring and education of inhalation
To investigate the effect of supervised nebulizer therapy | during study period (3 and 6 months)
  supervised nebulizer therapy
To correlate unobtrusive monitoring parameters and explore the feasibility and acceptance | during study period (3 and 6 months)
  unobtrusive monitoring parameters
To assess the perception of dyspnea in children | during study period (3 and 6 months)
  perception of dyspnea
To analyze the preluding period before an asthma exacerbation | during study period (3 and 6 months)
  preluding period
To identify the patient characteristics of children with successful eHealth care outcomes | during study period (3 and 6 months)
  patient characteristics

CONTACTS AND LOCATIONS:
Overall Officials: B.J. Thio, Pediatrician, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- MST, Enschede, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Kamp M, Hengeveld V, Willard N, Thio B, de Graaf P, Geven I, Tabak M. Remote Patient Monitoring and Teleconsultation to Improve Health Outcomes and Reduce Health Care Utilization of Pediatric Asthma (ALPACA Study): Protocol for a Randomized Controlled Effectiveness Trial. JMIR Res Protoc. 2023 Jul 3;12:e45585. doi: 10.2196/45585. PMID 37399066